CLINICAL TRIAL: NCT00235794
Title: An Open Label Study of Exploratory Pharmacogenomics and Pharmacologic Effects of Neoadjuvant Oral Temsirolimus in Newly Diagnosed Prostate Cancer Patients Undergoing Radical Prostatectomy Who Have a High Risk of Relapse
Brief Title: An Open Label Exploratory Study in Newly Diagnosed Prostate Cancer Patients
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Wyeth is now a wholly owned subsidiary of Pfizer (Industry)
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: 3066A1-132
Record Dates: First submitted 2005-10-06; First posted 2005-10-10 (Estimated); Last update posted 2007-12-27 (Estimated); Status verified 2007-12

CONDITIONS: Prostatic Neoplasms
MeSH Terms: conditions — Prostatic Neoplasms | interventions — temsirolimus

INTERVENTIONS:
Drug: temsirolimus

SUMMARY:
Open-label exloratory pharmacodynamic and pharmacogenomic study to evaluate teh biologic effects of 3 dose levels (1mg, 5 mg, and 15 mg) of temsirolimus administered orally once daily for approximately 4 weeks (+/- 2 weeks) before prostatectomy

ELIGIBILITY:
Inclusion criteria:

* Histologically confirmed diagnosis of adenocarcinoma of the prostate gland via a minimum of 6 core biopsy samples.
* Subjects must be a candidate for radical prostatectomy
* No evidence of metastatic disease as determined by CT scans and bone scans

  * More criteria apply

Exclusion Criteria:

* Subjects from whom sufficient diagnostic biopsy material is not available for full characterization of the tumor
* Active Infection requiring antibiotic therapy, or serious intercurrent illness, active bleeding, or ongoing urinary tract infection necessitating rapid or emergent surgical resection
* Subjects who have had hormonal injection or implants which will last longer than 6 months

  * More criteria apply

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2004-01; Study Completion 2007-09 (Actual)

PRIMARY OUTCOMES:
To determine the effects of oral temsirolimus on changes in phosphorylation state of proteins in the mTOR signaling pathway in tumor tissue and on phosphorylation state of mTOR pathway proteins and on global and targeted gene expression pattern PBMCs

SECONDARY OUTCOMES:
Determine effects of oral temsirolimus on global and targeted gene expression; compare effects in the tumor and PBMCs; obtain preliminary information on potential antitumor effects; evaluate PK using whole blood and tumor tissue.
To evaluate the relationship between PTEN status and the pharmacodynamic/pharmacogenomic effects of temsirolimus and to determine the effects of temsirolimus on changes in protein expression patterns in the plasma

CONTACTS AND LOCATIONS:
Overall Officials: Medical Monitor, Study Director — Wyeth is now a wholly owned subsidiary of Pfizer
Locations (1):
- Houston, Texas, United States